CLINICAL TRIAL: NCT06948708
Title: The Predictive Role of Heart Rate Variability in Postoperative Nausea and Vomiting Among Female Patients Undergoing Elective Laparoscopic Cholecystectomy: A Prospective Observational Study
Brief Title: Predictive Role of HRV for PONV in Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mahmut Sami TUTAR, Associate Professor, Department of Anesthesiology and Reanimation, Konya City Hospital
Other Study IDs: 10.04.2025/ 04-604-02
Record Dates: First submitted 2025-04-15; First posted 2025-04-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Nausea and Vomiting (PONV); Heart Rate Variability (HRV); Laparoscopic Cholecystectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients who develop postoperative nausea and/or vomiting within the first 24 hours after laparoscopic cholecystectomy.
- 2: Patients who do not experience postoperative nausea or vomiting within the first 24 hours after laparoscopic cholecystectomy.

SUMMARY:
Postoperative nausea and vomiting (PONV) are among the most common complications following general anesthesia (GA), significantly affecting patient comfort and recovery. Although various risk factors for PONV have been identified-such as female sex, non-smoking status, and history of motion sickness-these predictors are not always sufficient to determine individual risk accurately.

Heart rate variability (HRV) reflects autonomic nervous system (ANS) balance and has been proposed as a potential physiological biomarker for predicting PONV. Reduced HRV is associated with increased vagal imbalance, which may contribute to gastrointestinal (GI) dysregulation and PONV.

This prospective observational study aims to investigate the predictive value of HRV in estimating the incidence and severity of PONV in female patients undergoing elective laparoscopic cholecystectomy (LC). A total of 110 participants will be enrolled, and preoperative and early postoperative HRV measurements will be obtained using a validated chest-strap heart rate monitor (Polar H10). HRV parameters, including the standard deviation of normal-to-normal intervals (SDNN), the root mean square of successive differences (RMSSD), and the low-frequency/high-frequency (LF/HF) ratio, will be analyzed via the Elite HRV application. Standardized anesthesia, analgesia, and antiemetic protocols will be used for all participants. PONV severity will be assessed over the first 24 hours postoperatively using a 4-point scale.

The primary objective is to evaluate whether preoperative HRV can predict PONV occurrence. Secondary outcomes include correlations between HRV parameters and PONV severity.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 65 years
* Scheduled for elective laparoscopic cholecystectomy
* American Society of Anesthesiologists (ASA) physical status I
* Body mass index (BMI) < 35 kg/m²
* Non-smokers
* Able and willing to provide written informed consent

Exclusion Criteria:

* History of cardiovascular, neurological, or gastrointestinal disease
* Use of medications affecting HRV (e.g., antihypertensives, diuretics, atropine, antidepressants, antipsychotics, steroids)
* Presence of systemic diseases that may affect PONV risk
* Inability to comply with study procedures

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients aged 18-65 years, scheduled for elective laparoscopic cholecystectomy under general anesthesia at a tertiary care hospital.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Association between preoperative HRV and postoperative nausea and vomiting (PONV) within 24 hours | Within 24 hours postoperatively
  Preoperative HRV parameters (SDNN, RMSSD, LF/HF ratio) measured during a 5-min rest using Polar H10/Elite HRV. PONV assessed every 4 hours for 24 hours post-surgery using a 5-point ordinal scale (0-4). The predictive association between HRV and PONV incidence/severity will be evaluated.

SECONDARY OUTCOMES:
Preoperative HRV parameters (SDNN, RMSSD, LF/HF ratio). | Within 24 hours postoperatively
  Preoperative HRV parameters (SDNN, RMSSD, LF/HF) measured during a 5-min rest (Polar H10/Elite HRV). PONV assessed every 4 hours for 24 hours using a 5-point ordinal scale (0-4). Association between HRV and PONV incidence/severity will be evaluated.
Postoperative HRV parameters (SDNN, RMSSD, LF/HF ratio). | 1 hour postoperative (PACU).
  Postoperative HRV parameters (SDNN [ms], RMSSD [ms], LF/HF ratio) will be measured at the 1st postoperative hour in the PACU using the Polar H10 heart rate sensor and analyzed via the Elite HRV application. These values will be compared to preoperative measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional policies and data privacy concerns.